CLINICAL TRIAL: NCT03502837
Title: Effects of Emotional Stimuli in Patients With Disorders of Consciousness: An Electroencephalography and Neuroimaging Study
Brief Title: Effects of Emotional Stimuli in Patients With Disorders of Consciousness
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: event-related potential
Record Dates: First submitted 2018-03-18; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2017-09

CONDITIONS: Disorder of Consciousness
Keywords: ERP;DOC;auditory
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: age-matched right-handed healthy volunteers
  Interventions: Other: emotional sound and neutral sound
- the mininally conscious state: Patients present reproducible signs of awareness such as purposeful eye movements or response to verbal order
  Interventions: Other: emotional sound and neutral sound
- the vegetative state: Patients preserved autonomous functioning (e.g., preserved sleep-wake cycles),but without awareness of oneself or of the environment
  Interventions: Other: emotional sound and neutral sound

INTERVENTIONS:
Other: emotional sound and neutral sound — Neutral voice is a meaningless sound (namely the interjection "ah") and the emotional stimuli were the same voice pronouncing the same word with an emotional prosody of happiness or sadness.The stimulus material consisted of positive and negative sound selected from the International Affective Digitalized Sounds (IADS) database.In order to identify experimental stimuli sets that were matched for ratings of arousal and valence between the two valence types,investigators used an algorithm to equate normative valence and arousal ratings for the selection of auditory stimuli.

SUMMARY:
Disentangling the vegetative state from the minimally conscious state is often difficult when relying only on behavioral observation. In this study, the investigators explored a new event-related potential paradigm as an alternative method for the detection of voluntary brain activity and cognitive abilities in the patients with disorders of consciousness.

DETAILED DESCRIPTION:
Auditory emotional stimuli have potential beneficial effects on cognitive functions and consciousness in patients with disorders of consciousness (DOC); however, precise and accurate quantitative indices to estimate cerebral activation to different auditory stimuli remain scarce. In this study, investigators assessed the response of different brain regions to emotional stimuli using ERP(Event-related potential),and further investigated the brain activation network.

ELIGIBILITY:
Patients:

Inclusion Criteria:

1. Disorders of consciousness (Traumatic brain injury, stroke or anoxic encephalopathy)
2. Coma diagnosis (Plum and Posner, 1966), vegetative state (Task Force, 1994) or minimally conscious state (Giacino, Ashwal et al. 2002)
3. Lack of autonomic crisis since one week minimum
4. Medical condition considered stable
5. Patients who do not present hearing loss. Peaks I and II of Brainstem Auditory Evoked Potentials (BAEP) will be normal.

Exclusion Criteria:

1. hearing Problem
2. Uncontrolled Epilepsy
3. Autonomic crises
4. Medical unstable state
5. Pregnant or likely to be (interrogation data) or breastfeeding woman

Healthy controls:

Inclusion Criteria:

1. Subjects with normal hearing
2. Absence of neurological disorder
3. Subjects able to understand the experimental instructions

Exclusion Criteria:

1. Hearing problems and / or hearing loss higher than 30 decibels Hearing Level (dB HL) at a frequency band from 250 to 8000 Hz
2. Neurological disorders
3. Pregnant or likely to be (interrogation data) or breastfeeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy controls and 30 patients in dicorders of consciousness(15 VS and 15 MCS)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
electrophysiological index:the cognitive event-related potentional components | from 200 msec before the stimuli onset to 1000ms after the auditory stimulation
  The event-related potential waveforms uncover voluntary responses to external stimuli that could assist in detecting signs of consciousness to reduce the risk of misdiagnosis. P300 is a large positive going potential that increases in amplitude from the frontal to parietal electrodes and has a peak latency of about 300 ms for auditory and 400 ms for visual stimuli. And N1 is a negative potential in the posterior superior temporal lobe with the peak latency of about 170ms.Peak amplitudes and latency were obtained for the interest ERP components(N1,P300) .Peak amplitudes and latency for were analysed in a series of repeated-measures ANOVAs for each component (N1, P2), with factors of condition (emotion: mean happy/angry vs. neutral).

SECONDARY OUTCOMES:
CRS-R(Coma Recovery Scale-Revised) | 30 minutes before the auditory stimualtion and 30 minutes after each stimulation
  CRS-R has been designed to differentiate VS from MCS and consists of 23 hierarchically arranged items that comprise six subscales addressing arousal, auditory, visual, motor, oromotor/verbal, and communication functions. The lowest item on each subscale represents reflexive activity while the highest item represents cognitively mediated behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No